CLINICAL TRIAL: NCT01894581
Title: Effects of Dietary Omega-3 Fatty Acids on Reproductive Hormones in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-1420; U54HD058155-05 (NIH)
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2016-07-13 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Obesity; Fertility
MeSH Terms: conditions — Obesity | interventions — Omacor; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese Women (Experimental): Women with a BMI of greater than or equal to 30 kg/m2 underwent all study interventions, including taking 5 g daily of LOVAZA. Women underwent 8 hours of frequent blood sampling every 10 minutes both at baseline and after LOVAZA supplementation. Each frequent blood sampling included IV administration of GnRH at 6 hours.
  Interventions: Dietary Supplement: LOVAZA; Drug: GnRH
- Normal Weight (Active Comparator): Women with a BMI of between 18-25 kg/m2 underwent all study interventions, including taking 5 g daily of LOVAZA for one cycle. Women underwent 8 hours of frequent blood sampling every 10 minutes both at baseline and after LOVAZA supplementation. Each frequent blood sampling included IV administration of GnRH at 6 hours.
  Interventions: Dietary Supplement: LOVAZA; Drug: GnRH

INTERVENTIONS:
Dietary Supplement: LOVAZA — Subjects will be instructed to take 2 grams twice daily of oral omega-3-acid ethyl esters (Lovaza) starting with day 1 to 3 of their menstrual period. Each capsule contains 60mg of other omega-3 FA. On day 1 of their subsequent menstrual period, subjects will be instructed to discontinue.
  Other Names: Omega-3-acid ethyl esters
Drug: GnRH — An intravenous bolus of exogenous GnRH (75 ng/kg dosing based on total body weight) will be administered at 6 hours.
  Other Names: Gonadorelin (GnRH)

SUMMARY:
The United States has the highest prevalence of obesity among all countries surveyed in 2012 by the Organization for Economic Cooperation and Development. Maternal obesity is linked with anovulation, menstrual cycle abnormalities, subfertility, fetal loss, obstetrical complications and congenital anomalies. Changes in reproductive hormones and diminished oocyte quality have also been demonstrated. A gap of knowledge exists as the mechanisms underlying these harmful effects are poorly understood and no specific treatments exist.

This proposal will test the hypothesis that dietary omega-3 fatty acids (FA) will improve the output of hypothalamicpituitary- ovarian axis in obese women. The investigators will perform paired assessments before and after supplementation in 10 obese and 10 normal weight women. To test the pituitary and hypothalamic output, the investigators will examine the luteinizing hormone (LH) and follicle-stimulating hormone (FSH) responsiveness during frequent blood sampling. To test the corpus luteum function, the investigators will examine urinary reproductive hormones (E1c, estrone conjugates, and pregnanediol glucuronide (Pdg)) over an entire menstrual cycle. The investigators ultimate goal is to collect preliminary data for an adequately powered randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-42 at study entry
2. Regular menstrual cycles every 25-40 days
3. BMI at least 30 kg/m2 (obese) or between 18.5 and 25 kg/m2 (normal)
4. Good general health
5. Prolactin and thyroid-stimulating hormone (TSH) within normal laboratory ranges at screening, baseline hemoglobin >11 gm/dl.

Exclusion Criteria:

1. Diagnosis of polycystic ovary syndrome (by ultrasound or hyperandrogenic symptoms)
2. Fish or seafood allergy or hypersensitivity (e.g., anaphylactic reaction) to omega-3-acid ethyl esters or any component of the formulation
3. Coagulopathy or receiving therapeutic anticoagulation (due to potential for interaction with omega-3 FA)
4. History of chronic disease affecting hormone production, metabolism or clearance (including diabetes mellitus)
5. Abnormal renal or liver function at screening
6. Current use of thiazolidinediones or metformin (known to interact with reproductive hormones)
7. Use of hormones affecting hypothalamic output (HPO) axis (such as hormonal contraceptives) within three months of entry
8. Strenuous exercise (>4 hours of intense physical activity per week)
9. Pregnancy
10. Breast-feeding
11. Current active attempts to conceive
12. History of significant recent weight loss or gain

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Polotsky, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Bauer JL, Kuhn K, Bradford AP, Al-Safi ZA, Harris MA, Eckel RH, Robledo CY, Malkhasyan A, Johnson J, Gee NR, Polotsky AJ. Reduction in FSH Throughout the Menstrual Cycle After Omega-3 Fatty Acid Supplementation in Young Normal Weight but not Obese Women. Reprod Sci. 2019 Aug;26(8):1025-1033. doi: 10.1177/1933719119828099. Epub 2019 Feb 17. PMID 30773100
- [Derived] Al-Safi ZA, Liu H, Carlson NE, Chosich J, Harris M, Bradford AP, Robledo C, Eckel RH, Polotsky AJ. Omega-3 Fatty Acid Supplementation Lowers Serum FSH in Normal Weight But Not Obese Women. J Clin Endocrinol Metab. 2016 Jan;101(1):324-33. doi: 10.1210/jc.2015-2913. Epub 2015 Nov 2. PMID 26523525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 regularly menstruating obese and normal-weight women were recruited from the community through campus-wide advertisements.
Pre-assignment Details: Potential participants were screened out if they had polycystic ovary syndrome, allergies to seafood, used medications known to affect reproductive hormones, used exogenous sex steroids within the last 3 months, exercised vigorously more than 4 hours weekly, or were attempting pregnancy. Eligible subjects then had a baseline physical examination.
Groups:
- Obese: BMI >= 30 kg/m2
- Normal Weight: BMI 18-25 kg/m2
Period: Overall Study
Arm/Group | Obese | Normal Weight
Started | 20 | 19
Completed | 15 | 12
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Screen Failure | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese | Normal Weight | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (1.2) | 28.4 (1.2) | 31.6 (5.3)
Sex/Gender, Customized [Number; unit: participants]
  Female | 15 | 12 | 27
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 27
BMI [Mean (Standard Deviation); unit: kg/m^2] | 37.8 (1.5) | 21.8 (.5) | 31.6 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Average LH Pulse Amplitude
Description: To test the pituitary and hypothalamic output, we examined LH secretion (unstimulated and in response to gonadotropin-releasing hormone (GnRH) stimulation) during 8-hour blood sampling studies at 10 min intervals. The primary outcome measure is the change in the average LH pulse amplitude for each patient from baseline to after supplementation.
Time Frame: 10 minute intervals during 8 hour blood sampling studies. Subjects will undergo two menstrual cycles of study, one prior to dietary supplementation and one after supplementation.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Obese | Normal Weight
Number analyzed (Participants) | 15 | 12
IU/L | -.04 (.2) | .4 (.4)

ADVERSE EVENTS:
Time Frame: During approximately one menstrual cycle.
Description: Adverse event data were collected for the duration of the participant's participation, which was approximately one menstrual cycle. Data were from all subjects were collected from June of 2013 to February of 2015.
Arm/Group | Obese | Normal Weight
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 0/15 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No